CLINICAL TRIAL: NCT01212289
Title: The Use of Rotational Thromboelastometry ROTEM® to Characterize Coagulation Abnormalities in Pediatric Cardiac Surgical Patients: A Prospective Pilot Study
Brief Title: Use of ROTEM® in Pediatric Cardiac Surgical Patients
Acronym: PedsROTEM
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1005011027
Record Dates: First submitted 2010-09-24; First posted 2010-09-30 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Congenital Heart Defect
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For each group, a small amount of blood will be obtained for ROTEM® analysis after induction of anesthesia but before skin incision and again following cardiopulmonary bypass, 5 minutes following protamine administration.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary cardiac surgery: Pediatric patients receiving primary cardiac surgery
- Reoperation: Pediatric patients receiving cardiac surgery reoperation

SUMMARY:
Cardiac surgery requiring use of a heart-lung machine, also known as cardiopulmonary bypass (CPB) can induce abnormalities in blood coagulation (clotting) that lead to excessive blood loss during and after operation. While of significant concern in adults, this problem takes on even greater importance in children due to the simple fact that they have a smaller blood volume. It is well known that if a child has previously undergone a heart operation, they are at increased risk of bleeding should more cardiac surgery be required ("reoperation"). The processes regulating blood coagulation are extraordinarily complex, and little is known about the exact mechanisms that contribute to the increased bleeding associated with cardiac reoperation in children. Rotational thromboelastometry (ROTEM®) is a technology that can provide, at the bedside, detailed information about coagulation abnormalities. While not currently approved for general use in the United States, in Europe ROTEM® has been used to guide administration of the blood products in surgery based upon determination of specific coagulation abnormalities. Importantly, there is now evidence that guidelines for transfusion therapy based on ROTEM® reduce transfusion requirements thus decreasing patient exposure to blood products. Whether the use of ROTEM® has potential benefit for pediatric cardiac surgical patients has not been studied. Accordingly, the present study was designed to provide preliminary data comparing coagulation profiles between children undergoing cardiac reoperation to those having primary procedure.

The investigators hypothesize that ROTEM® analysis will detect a pattern of impaired coagulation in children undergoing reoperation. The overall objective of the four assays of ROTEM® analysis therefore, is to provide information that can be used to devise a rational transfusion protocol for pediatric cardiac surgical subjects.

DETAILED DESCRIPTION:
Specific aims of the proposed pilot studies are to:

1. Use bedside blood analysis with ROTEM® in pediatric cardiac surgical patients to provide preliminary information on the nature of coagulation abnormalities.
2. Compare ROTEM® coagulation profiles between subjects having primary surgery and those undergoing reoperation.

In order to test the study hypothesis, pediatric subjects scheduled to undergo cardiac surgery involving CPB will be recruited for two study groups: a) primary surgery; b) reoperation. For each group, a small amount of blood will be obtained for ROTEM® analysis after induction of anesthesia but before skin incision and again following Cardiopulmonary Bypass, 5 minutes after protamine administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital heart disease undergoing cardiac surgery needing cardiopulmonary bypass.
* Males and females
* Age 1 year to 6 years
* Informed consent obtained

Exclusion Criteria:

* Known pre-existing haemostatic abnormalities
* Emergency surgery
* Pre-operative treatment with prostaglandin infusion or any other medication known to interfere with platelet function or cause coagulation abnormalities .
* Inclusion in another clinical research study
* Refusal or inability of patient's parent to sign the Informed Consent Form in English.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minors from the ages 1-6 years old receiving cardiac surgery using a cardiopulmonary bypass machine
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2010-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To obtain pre- and post-cardiopulmonary bypass (CPB) coagulation profiles using ROTEM® in pediatric patients undergoing cardiac surgery with CPB | Profiles will be collected after induction of anesthesia and before CPB, and after CPB, 5 minutes after protamine adminsitration
  A small blood sample from an already existing arterial line will be taken from the patient at these times and analyzed using the ROTEM® machine.

SECONDARY OUTCOMES:
To compare ROTEM® coagulation profiles between subjects having primary surgery and those having a reoperation | 1.3 years

CONTACTS AND LOCATIONS:
Overall Officials: Aarti Sharma, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital/ Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Background] Haizinger B, Gombotz H, Rehak P, Geiselseder G, Mair R. Activated thrombelastogram in neonates and infants with complex congenital heart disease in comparison with healthy children. Br J Anaesth. 2006 Oct;97(4):545-52. doi: 10.1093/bja/ael206. Epub 2006 Jul 27. PMID 16873390
- [Background] Osthaus WA, Boethig D, Johanning K, Rahe-Meyer N, Theilmeier G, Breymann T, Suempelmann R. Whole blood coagulation measured by modified thrombelastography (ROTEM) is impaired in infants with congenital heart diseases. Blood Coagul Fibrinolysis. 2008 Apr;19(3):220-5. doi: 10.1097/MBC.0b013e3282f54532. PMID 18388502
- [Background] Straub A, Schiebold D, Wendel HP, Hamilton C, Wagner T, Schmid E, Dietz K, Ziemer G. Using reagent-supported thromboelastometry (ROTEM) to monitor haemostatic changes in congenital heart surgery employing deep hypothermic circulatory arrest. Eur J Cardiothorac Surg. 2008 Sep;34(3):641-7. doi: 10.1016/j.ejcts.2008.05.028. Epub 2008 Jun 25. PMID 18579398
- [Background] Segal JB, Dzik WH; Transfusion Medicine/Hemostasis Clinical Trials Network. Paucity of studies to support that abnormal coagulation test results predict bleeding in the setting of invasive procedures: an evidence-based review. Transfusion. 2005 Sep;45(9):1413-25. doi: 10.1111/j.1537-2995.2005.00546.x. PMID 16131373
- [Background] Spalding GJ, Hartrumpf M, Sierig T, Oesberg N, Kirschke CG, Albes JM. Cost reduction of perioperative coagulation management in cardiac surgery: value of "bedside" thrombelastography (ROTEM). Eur J Cardiothorac Surg. 2007 Jun;31(6):1052-7. doi: 10.1016/j.ejcts.2007.02.022. Epub 2007 Mar 29. PMID 17398108